CLINICAL TRIAL: NCT02191670
Title: A Post-registration, Open Label Therapeutic Observational Study of METALYSE® in Patients With Acute Myocardial Infarction In Russian Federation.
Brief Title: Observational Study of METALYSE® in Patients With Acute Myocardial Infarction In Russian Federation
Status: Completed | Type: Observational
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Other Study IDs: 1123.22
Record Dates: First submitted 2014-07-14; First posted 2014-07-16 (Estimated); Last update posted 2014-07-16 (Estimated); Status verified 2014-07

CONDITIONS: Myocardial Infarction
MeSH Terms: conditions — Myocardial Infarction | interventions — Tenecteplase

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- METALYSE®
  Interventions: Drug: METALYSE®

INTERVENTIONS:
Drug: METALYSE® — weight-adjusted dosage as single bolus over 5 to 10 seconds

SUMMARY:
Primary: To support the Regulatory Approval process of Metalyse® in Russian Federation. Secondary: To assess the efficacy and safety of single bolus of Metalyse® TNK-tissue plasminogen activator (TNK-tPA, Tenecteplase ) in patients with acute myocardial infarction in usual routine treatment after market launch

ELIGIBILITY:
Inclusion Criteria:

* onset of symptoms of AMI within 6 hours
* on a twelve-lead electrocardiogram (ECG), ST-segment elevation ≥ 0.1 millivolt (mV) in two or more limb leads, or > 0.2 mV in two or more contiguous precordial leads indicative of AMI, or left bundle-branch block
* age ≥ 18

Exclusion Criteria:

* significant bleeding disorder at present or within the past 6 months, known hemorrhagic diathesis
* patients with current concomitant oral anticoagulant therapy with International Normalised Ratio (INR) > 1.3
* any history of central nervous system damage (i.e. neoplasm, aneurysm, intracranial or spinal surgery)
* severe uncontrolled arterial hypertension (hypertension defined as blood pressure 180/110 mm Hg (systolic BP > 180 mm Hg and/or diastolic BP > 100 mm Hg) on one single reliable measurement during current admission prior to study enrolment
* major surgery, biopsy of a parenchymal organ, or significant trauma within the past 2 months (this includes any trauma associated with the current AMI), recent trauma to the head or cranium
* prolonged or traumatic cardiopulmonary resuscitation (> 2 minutes) within the past 2 weeks
* severe hepatic dysfunction, including hepatic failure, cirrhosis, portal hypertension (esophageal varices) and active hepatitis
* diabetic hemorrhagic retinopathy or other hemorrhagic ophthalmic conditions
* active peptic ulceration
* arterial aneurysm and known arterial/venous malformation
* neoplasm with increased bleeding risk
* Acute pericarditis and/or subacute bacterial endocarditis
* Acute pancreatitis
* hypersensitivity to the active substance tenecteplase and to any of the excipients
* use of Abciximab (ReoPro®) or other marketed GPIIb/IIIa antagonists within the preceding 12 hours
* any minor head trauma and any other trauma occurring after onset of the current myocardial infarction
* any known history of stroke or transient ischemic attack or dementia
* pregnancy or lactation, parturition within the previous 30 days. Women of childbearing potential must have a negative pregnancy test
* any known active participation in another investigative drug study or device protocol in the past 30 days
* previous enrollment in this study
* inability to follow protocol and comply with follow-up requirements
* any other condition that the investigator feels would place the patient at increased risk if the investigational therapy is initiated

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: primary care clinic
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2005-04; Primary Completion 2006-01 (Actual)

PRIMARY OUTCOMES:
Number of serious adverse events (SAE) | up to 30 days

SECONDARY OUTCOMES:
In-hospital rate of death | up to 30 days
In-hospital rate of stroke | up to 30 days
In-hospital rate of intracranial hemorrhage | up to 30 days
In-hospital rate of major bleeding | up to 30 days
In-hospital rate of non-fatal cardiac events | up to 30 days
Clinical benefit of routine use of Metalyse®, defined as the absence of 30- day mortality and in-hospital disabling stroke | up to 30 days